CLINICAL TRIAL: NCT04786028
Title: A Phase 2 Multi-Center, Open Label Study of Isatuximab Added to Standard CyBorD Induction and Lenalidomide Maintenance Treatments in Newly Diagnosed, Transplant Eligible Multiple Myeloma
Brief Title: A Study of Isatuximab Added to Standard CyBorD Induction and Lenalidomide Maintenance Treatments in ND-TEMM
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Canadian Myeloma Research Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMRG 008
Record Dates: First submitted 2021-01-22; First posted 2021-03-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Multiple Myeloma
Keywords: Hematologic Diseases; Neoplasms; Multiple Myeloma; Isatuximab; Cyclophosphamide; Dexamethasone; Bortezomib; Lenalidomide
MeSH Terms: conditions — Multiple Myeloma; Hematologic Diseases; Neoplasms | interventions — isatuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Isatuximab with CyBorD and Lenalidomide Maintenance (Experimental): This is a single arm study of Isatuximab administered intravenously in combination with cyclophosphamide, bortezomib and dexamethasone (CyBorD), and Lenalidomide maintenance treatment
  Interventions: Other: Isatuximab

INTERVENTIONS:
Other: Isatuximab — Brand name for interventional drug is Sarclisa

SUMMARY:
This is a phase II multi-center, open label, single arm study to evaluate the safety and efficacy of Isatuximab administered intravenously in combination with CyBorD induction treatment and Lenalidomide maintenance treatment in a 28-day long cycle in autologous stem cell transplant-eligible patients.

DETAILED DESCRIPTION:
This is a phase II, multicenter, open label, single arm study that will evaluate the safety and efficacy of Isatuximab administered intravenously at 10 mg/kg in combination with CyBorD induction treatment and Lenalidomide maintenance treatment in a 28-day long cycle in autologous stem cell transplant-eligible patients.

The induction treatment consists of four cycles of Isa-CyBorD. Isatuximab will be given on days 1, 8, 15 and 22 of cycle 1 and days 1 and 15 of cycle 2-4 in combination with Cyclophosphamide at 300 mg/m2 on days 1, 8, 15 and 22, Bortezomib at 1.5 mg/m2 on days 1, 8, 15 and 22 and Dexamethasone at 40 mg on days 1, 8, 15 and 22 of each 28-day cycle.

Following the induction phase, all subjects achieving at least stable disease will have stem cell mobilization per standard institutional procedures. This is followed by high dose chemotherapy (Melphalan 200 mg/m2) and autologous stem cell transplantation.

((If, for unexpected logistical reason, there is a foreseen delay of stem cell mobilization or transplantation of more than eight weeks after the end of cycle four of induction, an additional cycle of Isa-CyBorD can be given at the investigator's discretion.))

The maintenance treatment consisting of Isatuximab at 10 mg/kg administered intravenously on days 1, 8, 15 and 22 of cycle 1, days 1 and 15 of cycle 2 and 3 and day 1 all subsequent 28-day maintenance cycles in combination with Lenalidomide administered orally at 10 mg on days 1-21 of each 28-day cycle will be administered starting at day 100 (+/- 7 days) after the transplant. Lenalidomide, if tolerated well, will be increased to 15 mg starting with cycle 3.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria to be eligible for participation in this study:

1. Males or females, age 18 to 75 years of age.
2. ECOG performance status score of 0, 1 or 2.
3. Life expectancy of at least 9 months
4. Measurable disease according to the IMWG criteria defined as

   1. Serum monoclonal paraprotein (M-protein) ≥ 10 g/L (if IgG) or ≥5g/L (if IgA, D, E or M)
   2. Urine M-protein ≥ 200 mg/24 h
   3. Serum free light chains (FLC) assay: Involved FLC level ≥ 100 mg/L and an abnormal serum free light chain ratio (< 0.26 or > 1 .65) if no M-protein detected in serum or urine
5. Newly Diagnosed Symptomatic Multiple Myeloma by IMWG criteria
6. The following laboratory results must be met within 10 days of first study drug administration:

   1. ANC ≥ 1.0 x 109/L
   2. Hemoglobin ≥ 80 g/L (transfusions permitted)
   3. Platelets ≥ 70 x 109/L (or ≥50 x 109/L if ≥50% plasmacytosis in bone marrow.
   4. Calculated CrCl ≥ 30 mL/min
   5. AST and ALT ≤ 3.0 x ULN
   6. Total bilirubin ≤ 2 x ULN unless known to have Gilbert's disease
   7. Corrected serum calcium ≤ 3.5 mmol/L
7. Have signed the informed consent documents indicating that the subject understands the purpose of and procedures required for the study and is willing to participate and adhere to the study protocol.
8. Females with child-bearing potential (FCBP) must agree to use 2 reliable forms of contraception* simultaneously or practice complete abstinence from heterosexual contact for at least 28 days before starting study drug, while participating in the study (including during dose interruptions), and for at least 150 days after study treatment discontinuation.
9. Females must agree to abstain from breastfeeding during study participation and 150 days after study drug discontinuation.
10. Males must agree to use a latex condom during any sexual contact with FCBP while participating in the study and for 150 days following discontinuation from this study, even if he has undergone a successful vasectomy.
11. Males must also agree to refrain from donating semen or sperm during the treatment phase and for 150 days after discontinuation from this study treatment.
12. All subjects must agree to refrain from donating blood while on study therapy and for 28 days after discontinuation from this study treatment.

Females of childbearing potential (FCBP): a female of childbearing potential is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months).

* The two methods of birth control used may be selected from the following categories, but the two methods cannot be selected from any one category: barrier method: i.e., condom (male or female) or diaphragm with spermicide; hormonal: i.e., contraceptive pill, patch; intrauterine device (IUD); vasectomy; or tubal ligation.

Exclusion Criteria:

Subjects who meet any of the following exclusion criteria are not eligible for enrollment:

1. Prior exposure to Isatuximab (or other anti-CD38 monoclonal antibody)
2. Prior treatment for Multiple Myeloma (MM) with the exception of corticosteroids not exceeding a total dose specified below:
3. Subjects who have received steroids within 2 weeks prior to starting study treatment or who have not recovered from side effects of such therapy. Concomitant therapy medications that include corticosteroids are allowed if subject receive ≤10 mg of prednisone per day, or equivalent, as indicated for other medical conditions, or up to 100 mg of hydrocortisone as pre-medication for administration of certain medications or blood products prior to enrolment in this study.
4. Prior history of malignancies, other than MM, unless the subject has been free of the disease for 3 years or longer. Exceptions include the following:

   1. Basal or squamous cell carcinoma of the skin
   2. Carcinoma in situ of the cervix or breast
   3. Adenocarcinoma of the prostate (TNM stage of T1 a or T1 b)
5. Other concurrent severe and/or uncontrolled medical conditions (i.e. uncontrolled diabetes, active or uncontrolled infection, acute diffuse pulmonary disease, pericardial disease, uncontrolled thyroid dysfunction or uncontrolled severe arterial hypertension) including abnormal laboratory values, that could cause unacceptable safety risks or compromise compliance with the protocol
6. History of or current uncontrolled cardiovascular disease including:

   1. Unstable angina, myocardial infarction, or known congestive heart failure Class III/IV (Appendix 5) within the preceding 12 months
   2. Transient ischemic attack within the preceding 3 months, pulmonary embolism within the preceding 2 months.
   3. Any of the following: sustained ventricular tachycardia, ventricular fibrillation, Torsades de Pointes, cardiac arrest, Mobitz II second degree heart block or third-degree heart block; known presence of dilated, hypertrophic, or restrictive cardiomyopathy.
   4. QTc prolongation as confirmed by ECG assessment at screening (QTc >470 milliseconds).
   5. Poorly controlled severe arterial hypertension.
7. Women who are pregnant, breastfeeding or planning to become pregnant while enrolled in this study, or within 90 days after the last dose of study medications. Male subject who plans to father a child while enrolled in this study, within 90 days after the last dose of study medications.
8. Known HIV positivity or active infectious hepatitis B or C
9. Known allergies, hypersensitivity to mannitol, corticosteroids, monoclonal antibodies or human proteins, or their excipients (refer to the Isatuximab IB), or known sensitivity to mammalian-derived products, if not amenable to premedication with steroids, or H2 blockers that would prohibit further treatment with these agents.
10. Known CNS involvement, plasma cell leukemia or amyloidosis.
11. Subjects who are receiving any other investigational agent Any other condition that, in the Investigator's opinion, would contraindicate the patient's participation in the clinical study due to safety concerns or compliance with clinical study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2021-12-08 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Response rate (VGPR or better) defined by IMWG criteria | 100 days
  To determine the response rate (VGPR or better) defined by IMWG criteria at 100 days (+/- 7 days) after the autologous stem cell transplant (ASCT).

CONTACTS AND LOCATIONS:
Locations (7):
- Canada (7):
  - Cross Cancer Institute, Edmonton, Alberta
  - Nova Scotia Health - QEII Health Sciences Centre, Halifax, Nova Scotia
  - Hamilton Health Sciences Centre, Hamilton, Ontario
  - The Ottawa Hospital General Campus, Ottawa, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Center, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No